CLINICAL TRIAL: NCT04502485
Title: Reduce Patient Discomfort With Water Exchange Method During Upper Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yu-Hsi hsieh (Other)
Responsible Party: Sponsor-Investigator, Yu-Hsi hsieh, Dr., Dalin Tzu Chi General Hospital
Organization: Dalin Tzu Chi General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: A10801002
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Patients Undergoing Diagnostic EGD
Keywords: water exchange; upper endoscopy; discomfort

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric water exchange (Experimental): Air will be minimally insufflated to partially open the lumen and any residual fluid will be suctioned when the scope passes through the esophagus. Upon entering the fundus of the stomach the air button will be turned off. Air pocket and gastric fluids will be removed by suctioning. Distilled water, delivered by a 50-ml syringe in 10ml-to-20 ml increments, will be infused to dislodge debris and air bubbles adhering the gastric mucosa and open the lumen. The infused water will be removed to keep the lumen almost completely collapsed before the scope advance further. Air will be opened when the scope enter the prepylorus area where there is usually an air pocket. The scope will enter the duodenal bulb and 2nd portion of duodenum where withdrawal inspection will start.
  Interventions: Procedure: Gastric water exchange
- Traditional air insufflation (Active Comparator): Air will be minimally insufflated and residual fluid suctioned during the entire insertion process. Usually, no water will be infused to cleanse the mucosa until the withdrawal phase.
  Interventions: Procedure: traditional air insufflation

INTERVENTIONS:
Procedure: Gastric water exchange — Upon entering the fundus of the stomach the air button will be turned off. Air pocket and gastric fluids will be removed by suctioning. Distilled water, delivered by a 50-ml syringe in 10ml-to-20 ml increments, will be infused to dislodge debris and air bubbles adhering the gastric mucosa and open the lumen. The infused water will be removed to keep the lumen almost completely collapsed before the scope advance further.
  Arms: Gastric water exchange
Procedure: traditional air insufflation — Air will be minimally insufflated and residual fluid suctioned during the entire insertion process. Usually, no water will be infused to cleanse the mucosa until the withdrawal phase.
  Arms: Traditional air insufflation

SUMMARY:
The aim of the study was to evaluate the application of water exchange method to upper endoscopy. We hypothesize that water exchange during upper endoscopy could reduce patient discomfort. The primary outcome will be the patient discomfort score during upper endoscopy. The secondary outcomes will include cleanliness score, techniques adequacy score, findings of the EGD, and willing to repeat the procedure, as well as the patient and endoscopist satisfaction score with the method.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will include those anticipated to undergo EGD , aged 20 to 65 at the time of enrollment

Exclusion Criteria:

* a therapeutic EGD
* sedation with other agents
* American Society of Anesthesiology (ASA) risk Class 3 or higher, renal failure
* age less than 20 years or more than 65 years
* pregnancy
* refusal to provide written informed consent. All participants signed written informed consents

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Discomfort during the procedure | 5 minutes after the procedure
  A VAS discomfort score (0, no discomfort; 10, most discomfort) graded by the patient,

SECONDARY OUTCOMES:
patient satisfaction score | 5 minutes after the procedure
  A VAS score (0, not satisfied at all; 10, most satisfied) graded by the patient
mucosa cleanliness score | 1 minutes after the procedure
  1, no need for irrigation; 4, need more than 50 ml of water irrigation
technique adequacy score | 1 minutes after the procedure
  1, excellent; 6, very poor

CONTACTS AND LOCATIONS:
Locations (1):
- Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Chiayi City, Taiwan, Taiwan

REFERENCES:
- [Background] Abraham N, Barkun A, Larocque M, Fallone C, Mayrand S, Baffis V, Cohen A, Daly D, Daoud H, Joseph L. Predicting which patients can undergo upper endoscopy comfortably without conscious sedation. Gastrointest Endosc. 2002 Aug;56(2):180-9. doi: 10.1016/s0016-5107(02)70175-2. PMID 12145594
- [Background] Meining A, Semmler V, Kassem AM, Sander R, Frankenberger U, Burzin M, Reichenberger J, Bajbouj M, Prinz C, Schmid RM. The effect of sedation on the quality of upper gastrointestinal endoscopy: an investigator-blinded, randomized study comparing propofol with midazolam. Endoscopy. 2007 Apr;39(4):345-9. doi: 10.1055/s-2006-945195. Epub 2007 Feb 7. PMID 17285514